CLINICAL TRIAL: NCT03623971
Title: Validation of the Utility of a Universal Cataract Intelligence Platform
Brief Title: Validation of a Universal Cataract Intelligence Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Xidian University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCPMOH2018- China7
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Cataract; Artificial Intelligence
Keywords: Cataract; Artificial Intelligence; Medical Referral Pattern
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial Intelligence (Experimental): A universal diagnostic system. An artificial intelligence to make comprehensive evaluation and treatment decision of cataract.
  Interventions: Device: Cataract AI agent

INTERVENTIONS:
Device: Cataract AI agent — An artificial intelligence to make comprehensive evaluation and treatment decision of different types of cataracts.

SUMMARY:
This study established and validated a universal artificial intelligence (AI) platform for collaborative management of cataracts involving multi-level clinical scenarios and explored an AI-based medical referral pattern to improve collaborative efficiency and resource coverage.The datasets were labeled using a three-step strategy: (1) categorize slit lamp photographs into four separate capture modes; (2) diagnose each photograph as a normal lens, cataract or a postoperative eye; and (3) based on etiology and severity, further classify each diagnosed photograph for a management strategy of referral or follow-up. A deep residual convolutional neural network (CS-ResCNN) was used for the image classification task. Moreover, we integrated the cataract AI agent with a real-world multi-level referral pattern involving self-monitoring at home, primary healthcare, and specialized hospital services.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent ophthalmic examination of the eye and recorded their ocular information in the primary healthcare center.

Exclusion Criteria:

The patients who cannot cooperate with the examinations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the cataract AI agent | 6 months
  AUC: area under the receiver operating curve; accuracy (ACC) = (TP + TN) / (TP + TN + FP + FN); sensitivity (SEN) = TP / (TP + FN); specificity (SPE) = TN / (TN + FP); TP = true positive; TN = true negative; FP = false positive; FN = false negative.